CLINICAL TRIAL: NCT06525051
Title: Examination of the Effect of Handhaler Tiotropium, a Long-acting Anticholinergic, on Anterior Chamber Parameters
Brief Title: Effect of Tiotropium on Eye Findings in the Treatment of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Hayriye Bektaş, Assistant Professor, Giresun University
Other Study IDs: GiresunU-PULMONOLOGY-HB-01
Record Dates: First submitted 2024-07-21; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Glaucoma, Angle-Closure
Keywords: COPD; Eye findings; Tiotropium; Intraocular pressure; Glaucoma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Glaucoma, Angle-Closure; Eye Manifestations; Glaucoma | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 consisted of COPD patients not receiving any treatment ( inhaled and/or systemic steroids, long-acting inhaled beta-2 agonists alone, theophylline and combined long-acting beta-2 agonists and long-acting anticholinergic ). These patients are early stage COPD patients.
- Group 2: Group 2 consisted of healthy volunteers for similar age and gender.
- Group 3: Group 3 consisted of COPD patients of the same age and gender with receiving only handhaler Tiotropium 18 mcg for three months.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — Tiotropium is a long-acting anticholinergic agent and has a bronchodilator effect. According to the COPD Gold 2024 guideline, it is one of the long-acting bronchodilator drugs used as the first choice in the treatment of group A COPD patients.
  Groups: Group 3

SUMMARY:
This study aimed to examine the effect of Tiotropium, which is used in the treatment of COPD, on eye symptoms.The study was conducted prospectively. Patients were examined in three groups. Thirty-six patients were included in each group in the study. Anterior chamber parameters, intraocular pressure values, and photopic-mesopic pupil diameters were measured at the initial visit for Group 1 and Group 2 patients, and at the third month of treatment for Group 3 patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a persistent, chronic inflammatory disease of the lungs. Tiotropium, used in the treatment of COPD, is a muscarinic receptor antagonist that provides long-acting bronchodilation. In this study the researchers aimed to investigate the effects of Tiotropium on eye anterior chamber parameters.

The study was conducted prospectively between October 2023 and April 2024 after obtaining local Ethics Committee approval (Giresun EAH KEAK 2023/180 and 9.10.2023/02). Patients diagnosed with COPD and included in Group A according to the GOLD 2024 guidelines, along with healthy volunteers, were enrolled. Patients diagnosed with COPD, with mMRC scale 0-1, CAT score <10, who had never experienced an exacerbation before or had a mild severity exacerbation once that not required hospitalization were considered as Group A. Patients were examined in three groups: Group 1 consisted of COPD patients not receiving treatment, Group 2 consisted of healthy volunteers for similar age and gender, and Group 3 consisted of COPD patients of the same age and gender with receiving Tiotropium 18 mcg Handihaler. A total of 108 patients, 36 patients in each group, were included in the study. Anterior chamber parameters, intraocular pressure values and photopic-mesopic pupil diameters were measured at the initial visit for Group 1 and Group 2 patients, and at the third month of treatment for Group 3 patients.

Anterior segment optical coherence tomography (AS-OCT) was used to measure anterior chamber and angle parameters, corneal topography was utilized to assess anterior chamber depth, pupil diameter measurements in mesopic and photopic conditions, and intraocular pressure (IOP) was calculated using Goldmann applanation tonometry. Each patient underwent a comprehensive ophthalmic evaluation, including testing of best-corrected visual acuity, slit-lamp biomicroscopy, and fundoscopic examination.

Corneal topography (Topcon Aladdin Corneal Topography, Japan) was used to evaluate anterior chamber depth and pupil diameter in mesopic and photopic conditions. Pupil diameters measured with corneal topography were obtained by the same researcher, using the same device, at the same times of day and under similar lighting conditions.

Intraocular pressure was measured using Goldman Applanation tonometry. All measurements were conducted by the same researcher around 10 a.m., using the same tonometer device, without any manipulation or negligible manipulation of the eyelids. Applanation was performed by rotating the dial on the Goldman tonometer previously set to 10 mm Hg. The procedure was repeated after one minute. If the difference between the first and second readings was greater than 2 mm Hg, a third reading was performed. The average of the data obtained from two readings was taken, and if a third reading was needed, the median was used instead.

This study is the first research that investigate the effects of Tiotropium on anterior chamber parameters, pupil diameters, and intraocular pressure in COPD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of COPD
2. Not receiving any COPD treatment
3. Receiving only 18 mcg Tiotropium treatment
4. With written consent

Exclusion Criteria:

1. Patients under 18 years of age 2. Pregnant women 3. Without written consent 4. Receiving the following medications: 4a. Inhaled and/or systemic steroids 4b. Long-acting inhaled beta-2 agonists 4c. Combined long-acting beta-2 agonists and long-acting anticholinergics 4d. Topical medication

5. Patients with the following comorbidities 5a. Glaucoma 5b. Cataract 5c. Hypertension 5d. Diabetes Mellitus 5e. Patients had previously undergone eyelid, refractive, or intraocular surgery, those with corneal diseases altering the corneal surface

6. Patients receiving topical medications for chronic eye diseases 7. Patients receiving medications for diabetes mellitus 8. Patients receiving medications for hypertension 8. Patients those using contact lenses

Ages: 47 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups were formed for the study. Group 1 consisted of COPD patients not receiving treatment, Group 2 consisted of healthy volunteers for similar age and gender, and Group 3 consisted of COPD patients of the same age and gender with receiving handhaler Tiotropium 18 mcg. Anterior chamber parameters, intraocular pressure values and photopic-mesopic pupil diameters were measured at the initial visit for Group 1 and Group 2 patients, and at the third month of treatment for Group 3 patients.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Tiotropium causes narrowing of the eye angles and an increase in intraocular pressure and pupil diameters. | Measurements were made in the third month of Tiotropium treatment.
  Tiotropium 18 mcg is a long-acting anticholinergic drug used in the treatment of COPD. In patients diagnosed with COPD who do not receive any steroid treatment and who are not diagnosed with hypertension, glaucoma, diabetes mellitus, cataract and who have not undergone eye surgery and using only handhaler Tiotropium 18 microgram, a narrowing of the eye angles, an increase in photopic-mesopic pupil diameters and intraocular pressure were detected in the third month of treatment.

SECONDARY OUTCOMES:
Tiotropium did not cause acute angle-closure glaucoma in COPD patients. | Measurements were made in the third month of Tiotropium treatment.
  Tiotropium 18 mcg is a long-acting anticholinergic drug used in the treatment of COPD. In patients diagnosed with COPD ( who do not receive any steroid treatment and who are not diagnosed with hypertension, glaucoma, diabetes mellitus, cataract and who have not undergone eye surgery ) using only handhaler Tiotropium 18 microgram, open angle-closure glaucoma was not observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun Training and Research Hospital, Giresun, Gi̇resun, Turkey (Türkiye)

REFERENCES:
- [Derived] Aksoy HB, Koc H. Effect of Tiotropium on eye findings in the treatment of chronic obstructive pulmonary disease. BMC Pulm Med. 2024 Aug 28;24(1):418. doi: 10.1186/s12890-024-03240-1. PMID 39198799